CLINICAL TRIAL: NCT03602118
Title: A Randomized, Double-blind, Parallel Group, Phase 3 Study to Evaluate the Efficacy of Phenobarbital Sodium Injection for the Treatment of Neonatal Seizures
Brief Title: Study to Evaluate Phenobarbital Sodium Injection for the Treatment of Neonatal Seizures
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor withdrawing the subject IND
Sponsor: PharPoint Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1021.121.039.00
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Neonatal Seizure
Keywords: clinical seizures,
MeSH Terms: interventions — Phenobarbital

STUDY DESIGN:
Intervention Model Description: This is a 1:1 randomized, double-blind, parallel-group, Phase 3 study.
Who Masked: Care Provider, Investigator
Masking Description: All efforts will be made to blind the investigator and other key personnel of which dosage the participant was randomized to. Study drug will be dispensed by the pharmacy via a syringe to the investigator or their designee. The study medication label should only contain the protocol number, subject number and any other pertinent information. If after 1 hour following the completion of the study drug infusion, the seizure is not controlled with the initial loading dose, the patient will be considered a treatment failure in the primary efficacy analysis of this protocol/study. At this point, the blinding for the treating provider/investigator will be lifted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phenobarbital Sodium Injection 20 mg (Active Comparator): Once participants are deemed to be eligible for participation in the study and randomized to the lower dose they will be given a loading dose of phenobarbital 20 mg/kg administered intravenously over the course of 30 minutes.
  Interventions: Drug: Phenobarbital Sodium Injection
- Phenobarbital Sodium Injection 40 mg (Active Comparator): Once participants are deemed to be eligible for participation in the study and randomized to the higher dose they will be given a loading dose of phenobarbital 20 mg/kg administered intravenously over the course of 30 minutes. ministered intravenously over the course of 30 minutes.
  Interventions: Drug: Phenobarbital Sodium Injection

INTERVENTIONS:
Drug: Phenobarbital Sodium Injection — Phenobarbitone Inj, Phenobarbitone SOD, Phenobarbitone Sodium
  Other Names: Phenobarbital Sodium Injection 20 mg; Phenobarbital Sodium Injection 40 mg

SUMMARY:
This is a randomized, double-blind, parallel-group, Phase 3 study to evaluate the efficacy of the administration of phenobarbital Sodium Injection, United States Pharmacopeia, (USP), in participants who have suffered from a clinical seizure. As neonatal seizures can have long-term adverse effects, including death, placebo-controlled studies are not appropriate for this population. This study is designed to show phenobarbital is effective at preventing subsequent seizures by demonstrating greater efficacy at the higher (40 mg/kg) dose compared to the lower dose (20 mg/kg). It is important to note that, although phenobarbital is not approved for the treatment of neonatal seizures, it is commonly used for this indication and is considered the first-line therapy in the US and by the World Health Organization. The minimum recommended dose of phenobarbital used to treat neonatal seizures is 20 mg/kg. Therefore, the lower dose of phenobarbital used in this study is considered an "effective" dose for the treatment of neonatal seizures. The design of this study allows for assessment of the minimum recommended dose with the maximum recommended dose to show the increased efficacy of the high dose in various measures of reduction in seizures.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, Phase 3 study to evaluate the efficacy of the administration of Phenobarbital Sodium Injection, USP in participants who have suffered from a clinical seizure. As neonatal seizures can have long-term adverse effects, including death, placebo-controlled studies are not appropriate for this population. This study is designed to show phenobarbital is effective at preventing subsequent seizures by demonstrating greater efficacy at the higher (40 mg/kg) dose compared to the lower dose (20 mg/kg). It is important to note that, although phenobarbital is not approved for the treatment of neonatal seizures, it is commonly used for this indication and is considered the first-line therapy in the United States, (US), and by the World Health Organization. The minimum recommended dose of phenobarbital used to treat neonatal seizures is 20 mg/kg. Therefore, the lower dose of phenobarbital used in this study is considered an "effective" dose for the treatment of neonatal seizures. The design of this study allows for assessment of the minimum recommended dose with the maximum recommended dose to show the increased efficacy of the high dose in various measures of reduction in seizures.

Study participants undergoing electrographic or electroclinical seizures lasting 10 seconds or longer will be randomized in a 1:1 fashion between the 2 treatment arms. Participants will receive either a 20-mg/kg or 40-mg/kg loading dose of Phenobarbital Sodium Injection, USP upon confirmation that the seizure was not due to metabolic imbalances. Randomization of participants with hypoxic-ischemic encephalopathy, (HIE), will be stratified between the dosing groups. Participants will further be stratified by treatment group for pharmacokinetics, (PK), analysis timepoints due to the limitations on the number of pharmacokinetics, (PK), samples that can be taken from each patient. After cessation of seizures the participants will remain in the hospital for 24 hours for continuous monitoring by electroencephalogram, (EEG).

According to recommended dosing of phenobarbital, participants in the 20-mg/kg treatment arm in whom seizure activity does not resolve after the first dose (20 mg/kg) will be given phenobarbital in 10-mg/kg increments (each hour) until the seizure activity resolves, up to a maximum total dose of 40 mg/kg. If the seizure activity is still not resolved, participants will be given a second-line anticonvulsant. The second-line therapy given will be determined by the attending physician and recorded in the study documentation. Participants in the 40-mg/kg treatment arm in whom seizure activity does not resolve after the initial loading dose of phenobarbital will be given a second-line anticonvulsant. The second therapy given will be determined by the attending physician and recorded in the study documentation.

ELIGIBILITY:
Inclusion Criteria:

1. Parental informed consent
2. Infants born at ≥ 35 + 0/7 weeks gestational age AND age 0-28 days after birth
3. Has evidence of an electrographic seizure lasting at least 10 seconds
4. Undergoing continuous electroencephalogram, (EEG), monitoring, including infants with hypoxic-ischemic encephalopathy concurrently treated with hypothermic cooling

Exclusion Criteria:

1. If the seizures are solely due to a transient abnormality, easily correctable, and unlikely to recur (for example, transient electrolyte abnormalities)
2. If the infant has been diagnosed with or there is a strong suspicion of an inborn error of metabolism, significant brain malformation, or microcephaly (< 3rd percentile)
3. If the infant has been diagnosed with an intrauterine viral infection
4. If the infant is not expected to survive to discharge

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
A change in the number of seizures in neonatal infants after administration of phenobarbital sodium injection | The 24 hour period after the initial loading dose of pheonobarbital sodium injection is given.
  Once a neonate has been identified as having a seizure by electroencephalogram he/she will be randomized to one of two doses of phenobarbital sodium injection, (20 mg/kg or 40 mg/kg). The number of neonates in each group will be observed for the end of any further seizures, also verified by electroencephalogram. In addition to observing when all seizure activity ended after the initial loading dose, the number of infants requiring a second dose of phenobarbital or second-line anti-convulsant therapy to treat unresolved or subsequent seizures will be observed in each randomization group, (phenobarbital sodium injection 20mg/kg or 40mg/kg) following the initial loading dose.

IPD SHARING:
Plan to Share IPD: No